CLINICAL TRIAL: NCT01909505
Title: Comparison of Salivary Testosterone With Serum Free Testosterone Done by Equilibrium Dialysis.
Brief Title: Comparison of Salivary and Serum Free Testosterone in Normal and Hypogonadal Men
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Saliva Biomarkers, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Saliva Testosterone
Record Dates: First submitted 2013-07-24; First posted 2013-07-26 (Estimated); Last update posted 2013-07-26 (Estimated); Status verified 2013-07

CONDITIONS: Known Androgen Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normal Males: Males with normal levels of serum testosterone
- Hypogonadal males: Males known to have low levels of serum testosterone

SUMMARY:
Low testosterone is a common male problem. The diagnosis of low testosterone often requires blood sampling and expensive testing. We want to know if measuring saliva testosterone can be used in place of blood sampling. Study participants will be asked to provide samples of blood and saliva for the measurement of testosterone. These results may lead to the development of a saliva test for testosterone.

DETAILED DESCRIPTION:
Testosterone is required for normal male health that is known to decline in aging or other conditions. Physiologically active testosterone, also known as "free" testosterone, is present as a small percentage of the total blood level, mostly bound to sex hormone binding globulin and albumin. Estimation of serum free testosterone is difficult and costly, requiring equilibrium dialysis of a serum sample. These binding proteins are not normally present in saliva. It is hypothesized that the free fraction of testosterone in blood is in equilibrium with the extravascular space, notably saliva. The sponsor proposes to test this hypothesis by sampling saliva and serum and measuring testosterone. Serum free testosterone will be measured following equilibrium dialysis. To perform this study approximately 40 eugonadal and 20 hypogonadal males will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* Normal male subjects aged 20-65 years

Exclusion Criteria:

* Women Smokers, HIV positive, diabetes, hepatatis C positive, subjects currently taking testosterone who are unwilling to suspend use for teh duration of the trial, subjects taking aldactone or medicines that may interfere with the protocol

Ages: 20 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Forty normal males and 20 male subjects, 25 to 65 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-06 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
blood and saliva testosterone | 1 year
  Measures of blood and saliva testosterone

CONTACTS AND LOCATIONS:
Overall Officials: West T Moore, M.D., Principal Investigator — Georgetown University
Locations (2):
- United States (2):
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - John's Hopkins University Medical Center, Baltimore, Maryland